CLINICAL TRIAL: NCT06533592
Title: A Prospective Randomized Study to Evaluate the Effect of the Type of Conduit-duct Anastomosis Using the Single/continuous Suture Technique on the Postoperative Course in Patients Undergoing Liver Transplantation from a Deceased Donor.
Brief Title: The Effect of the Type of Conduit-duct Anastomosis Technique on the Postoperative Course in Patients Undergoing Liver Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/ABM/01/00017
Record Dates: First submitted 2024-07-09; First posted 2024-08-01 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-06

CONDITIONS: Liver Transplant; Complications; Bile Duct; Stricture, Postoperative; Bile Leak; Quality of Life
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous suture technique (Experimental): Biliary duct-to-duct anastomosis performed with continous suture technique
  Interventions: Procedure: Continous suture technique
- Interrupted suture (Active Comparator): Biliary duct-to-duct anastomosis performed with interrupted suture technique - control group
  Interventions: Procedure: Interrupted suture technique

INTERVENTIONS:
Procedure: Continous suture technique — Duct-to-duct anastomosis will be performed using continuous suture technique for study group
  Arms: Continuous suture technique
Procedure: Interrupted suture technique — Duct-to-duct anastomosis will be performed using an interrupted suture for control group,
  Arms: Interrupted suture

SUMMARY:
The main objective of the trial is to compare the effect of two end-to-end duct-to-duct anastomosis surgical techniques using the continuous suture method versus interrupted method (control group) on reducing the risk of bile leakages in the 90-day follow-up period after liver transplantation and other postoperative complications resulting from them i.e.: the occurrence of a critical stenosis in the duct-to-duct anastomosis within 90 days. In addition, as part of the research experiment, long-term biliary complications will be assessed, i.e. occurring over a period of more than 90 days (a 2-year observation period of patients was assumed).

As part of the trial 284 patients qualified for the procedure of liver transplantation from a deceased donor will be included, in whom end-to-end anastomosis of the bile ducts will be performed. After entering the study, patients will be randomized to one of the groups. In the group of 142 patients, duct-to-duct anastomosis will be performed using an interrupted suture (control group), and the remaining patients will be performed using the continuous suture technique.

The analysis will also include surgical complications, complications related to early and late graft function, retransplantation and overall survival.

Additionally the analyses an analysis of the impact of the occurrence of a biliary complication on the quality of life of patients after liver transplantation will be performed on the basis of the EORTC QLQ-C30 forms.

The period of observation of the patient after the procedure is planned for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* elective liver transplantation
* informed consent to participate in the study
* recipient bile duct diameter over 3mm
* donor bile duct diameter over 3mm

Exclusion Criteria:

* age below 18
* pregnancy
* living donor liver transplantation
* split-liver or reduced-size liver transplantation
* liver transplantation other than from brain death donor
* liver transplantation with hepaticojejunostomy
* patients undergoing re-transplantation
* multi-organ transplantation
* recipient bile duct diameter below 3mm
* donor bile duct diameter below 3mm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Bile leakage | 90 days post transplantation
  Defined as bilirubin concentration in the drain fluid at least 3 times the serum bilirubin concentration or as the need for radiologic or operative intervention resulting from biliary collections or bile peritonitis up to 90 days post transplantation

SECONDARY OUTCOMES:
Critical biliary stricture | 90 days post transplantation
  Defined as the need for radiologic, endoscopic or operative intervention resulting from increased serum bilirubin concentration
Other surgical complications | 90 days post transplantation
  Occurence of complication assessed in Clavien-Dindo scale
Long-term biliary complications | 2 years post transplantation
  Defined as occurence of biliary leak, biliary stricture, peripheral cholangiopathy, recurrent cholangitis between 90 days and 2 years post transplantation
Overall survival | 2 years post transplantation
Overall graft survival | 2 years post transplantation
Impact of the occurrence of a biliary complication on the quality of life of patients | 2 years post transplantation
  Evaluated with EORTC QLQ-C30 form

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General, Transplantation and Liver Surgery UCC MUW, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided